CLINICAL TRIAL: NCT07371000
Title: Early Detection of Overactive Bladder and Elimination of Negative Impact on Quality of Life
Brief Title: Early Detection of OAB and Elimination of Negative Impact on Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: General University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UZIS 2024/3
Record Dates: First submitted 2026-01-14; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Overactive Bladder (OAB)
Keywords: Overactive bladder; Screening; Telemedicine; Online screening tool
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OAB Screening Arm (Other): Participants matching all the inclusion & exclusion criteria will undergo a standardized screening process for the diagnosis of OAB. This process involves the use of an online screening self-testing tool, where the data from individual questionnaires specific to OAB diagnosis will be evaluated by a specialist.
  Interventions: Other: Standardized Screening Protocol

INTERVENTIONS:
Other: Standardized Screening Protocol — After completing the online screening tool (including validated questionnaires), selected participants are offered an appointment with a specialist who will perform a diagnosis, confirm or rule out OAB and set up adequate therapy according to recommended procedures.

SUMMARY:
Overactive bladder (OAB) is one of the most common health problems in the adult population. The goal of this project is to improve the awareness of the problem and to correctly refer the targeted persons to a specialist or a doctor. This will be provided by an online screening tool, designed as web platform and mobile application, where the data will be stored in respect to GDPR. People with a positive result from the online screening tool will be offered an examination by a specialist (gynaecologist, urogynaecologist, urologist) involved in the project. The specialist will have access to the results from the online screening tool - he/she will log into the web platform with a view of the participants profile. He/she will perform the diagnosis, confirm or refute the diagnosis and complement it with any further diagnostic tests and set the standard treatment.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is one of the most common health problems in the adult population (15-20% prevalence), with just under half of those affected seeking professional medical help. The goal of this project is to improve the awareness of the problem and to correctly refer the targeted participants to a specialist or a doctor who is knowledgeable about the problem and who will set up an adequate therapy.

A targeted PR campaign will direct those interested in joining the pilot screening project to a website with information about OAB and information about the pilot screening process. The web platform will also guide the user to create a secure user profile to participate in the project, where they will complete validated questionnaires related to OAB, necessary personal and family history data to optimize follow-up diagnosis during the in-person examination with a specialist, and a validated questionnaire measuring quality of life. After completing the online screening tool, the user will be offered a referral to a specialist in the vicinity. Participation in the online screening tool will be conditional on checking the online Consent to Participate box and Consent to Disclose Personal Data in accordance with GDPR.

People with a positive result from the online screening tool will be offered an examination by a specialist (gynaecologist, urogynaecologist, urologist) involved in the project. The specialist will have access to the results from the online screening tool - he/she will log into the web platform with a view of the participant's profile. He/she will perform the diagnosis, confirm or refute the diagnosis and complement it with any further diagnostic tests and set the standard treatment.

The data collected will be used to properly evaluate the pilot project in line with its objectives. An analysis of the problems and risks of the project with regard to the whole pilot screening process and a simplified cost evaluation will also be carried out.

ELIGIBILITY:
Inclusion criteria:

* Signed Consent to Participate in the Project and Consent to the Processing of Personal Data (online and paper format)
* Men and women over 18 years of age with increased urinary frequency (more than 7 times in 24 hours)

Optional inclusion criteria:

- Nycturia and/or urge incontinence.

Exclusion criteria:

* Unsigned Consent to Participate in the Project and Consent to the Processing of Personal Data.
* Current treatment of OAB, acute problems, suspicion of another disease causing OAB symptoms (haematuria, suspected bladder cancer, etc.)
* Inflammation of the lower urinary tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Pilot testing with 1,000 participants | From enrollment to the end of examination in 3 months
  Pilot testing of the procedure on a sample of 1,000 people who will undergo an online self-diagnostic screening tool and be examined by a urogynecologist/urologist.
Number of participants (completion of anonymous screening test) | from enrollment up to 1 week
  Number of participants who complete anonymous screening test based on three questions reffering to urology health
Percentage of people with suspected OAB who agreed to participate in a follow-up examination with specialist | From enrollment up to 3 months
Percentage of people with a specialist confirmed diagnosis of OAB at the face-to-face visit | Through study completion, an average of 6 months
Percentage of people who attended follow-up examination after 3 months | Through study completion, an average of 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaromír Mašata, Professor, Study Director — General University Hospital of Prague
Locations (20):
- Czechia (20):
  - Brno University Hospital, Brno
  - GYN-LINE, s.r.o., Brno
  - České Budějovice Hospital, České Budějovice
  - Hospital Hořovice, Hořovice
  - University Hospital Hradec Králové, Hradec Králové
  - Hospital Jablonec nad Nisou, Jablonec nad Nisou
  - AGYNO s.r.o., Karlovy Vary
  - Oblastní nemocnice Kolín a.s., Kolín
  - Olomouc University Hospital, Olomouc
  - GYNOVA s.r.o., Ostrava
  - Hospital AGEL Ostrava - Vítkovice a.s., Ostrava
  - University Hospital Ostrava, Ostrava
  - Gyncare Michael Švec s.r.o., Pilsen
  - Mulačova nemocnice, Pilsen
  - General University Hospital, Prague
  - GynUp! s.r.o., Prague
  - University Hospital Bulovka, Prague
  - University Thomayer Hospital, Prague
  - Uroklinikum s.r.o., Prague
  - Sokolov Hospital, Sokolov